CLINICAL TRIAL: NCT05871619
Title: Clinical Efficacy of Combined Application of Diode Laser and Different Remineralizing Agents on Combined Application of Diode Laser and Different Remineralizing Agents on White Spot Lesions
Brief Title: Combined Application of Diode Laser and Different Remineralizing Agents on White Spot Lesions
Acronym: Whitespot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Amani abdullah Omar bin shahna, operative clinic, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P-OP-19-05
Record Dates: First submitted 2023-05-13; First posted 2023-05-23 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: White Spot Lesion of Tooth
Keywords: white spot lesion, diode laser, vita easy shade V

STUDY DESIGN:
Intervention Model Description: * The first group (A1B1):15 teeth with WSL were treated with Remin Pro with laser application.
  * The second group (A1B2): The contralateral 15 teeth were treated with Remin Pro without laser application.
  The third group (A2B1): 15 teeth with WSL were treated with X Pur Remin with laser application.
  * The fourth group (A2B2): The contralateral 15 teeth will be treated with XPur Remin without laser application.
  * The fifth group (A3B1): 15 teeth with WSL were treated with 5% sodium fluoride varnish with laser application.
  * The sixth group (A3B2): The contralateral 15 teeth were treated with 5% sodium fluoride without laser application
Who Masked: Investigator
Masking Description: To avoid bias and for proper randomization, the study will be done per patient using tossing a coin to assign the tooth to be either treated with Nano hydroxyapatite with fluoride or Nano hydroxyapatite with xylitol or sodium fluoride.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Remin Pro with laser application (Experimental): A photosensitizing-remineralizing agent mixture was prepared by adding pre-green dye (0.05ml) to 1 mg of the assigned remineralizing agents. The diode laser was irradiated immediately with Average power of 1 W, Exposure time of 10 s, diode 810 nm, continuous and non-contact mode, and Irradiation speed of 1mm/ sec.
  Interventions: Procedure: Remin Pro
- Remin pro without laser application (Experimental): Used a pea-sized amount with a brush and allowed it to remain on the teeth for at least three minutes as it was recommended by the manufacturer. Instructed the patient to avoid rinsing, eating, and drinking for 30 minutes
  Interventions: Procedure: Remin Pro
- Xpur remin with laser application (Experimental): A photosensitizing-remineralizing agent mixture was prepared by adding pre-green dye (0.05ml) to 1 mg of the assigned remineralizing agents. The diode laser was irradiated immediately with Average power of 1 W, Exposure time of 10 s, diode 810 nm, continuous and non-contact mode, and Irradiation speed of 1mm/ sec.
  Interventions: Procedure: X Pur Remin
- Xpur remin without laser application (Experimental): used a thin film of toothpaste on a micro brush and then applied it on the tooth surface for three minutes 2- Do not eat, drink or rinse for 30 minutes
  Interventions: Procedure: X Pur Remin
- fluoride varinsh with laser application (Experimental): A photosensitizing-remineralizing agent mixture was prepared by adding pre-green dye (0.05ml) to 1 mg of the assigned remineralizing agents. The diode laser was irradiated immediately with Average power of 1 W, Exposure time of 10 s, diode 810 nm, continuous and non-contact mode, and Irradiation speed of 1mm/ sec.
  Interventions: Procedure: Fluoride varnish
- fluoride varnish without laser application (Experimental): Used brush applicator to uniformly apply fluoride Varnish, covering the surface to be treated as a thin film.Instructed patient to avoid hard food, alcohol, brushing or flossing for the next 4
  Interventions: Procedure: Fluoride varnish

INTERVENTIONS:
Procedure: Remin Pro — A photosensitizing-remineralizing agent mixture was prepared by adding pre-green dye The diode laser was irradiated immediately with 1 W, Exposure time of 10 s, 810 nm, continuous and non-contact mode.
  Other Names: Experimental: Remin Pro with laser application; Experimental: Remin pro without laser application
  Arms: Remin Pro with laser application; Remin pro without laser application
Procedure: X Pur Remin — A photosensitizing-remineralizing agent mixture was prepared by adding pre-green dye The diode laser was irradiated immediately with 1 W, Exposure time of 10 s, 810 nm, continuous and non-contact mode.
  Other Names: Experimental: Xpur remin with laser application; Experimental: Xpur remin without laser application
  Arms: Xpur remin with laser application; Xpur remin without laser application
Procedure: Fluoride varnish — A photosensitizing-remineralizing agent mixture was prepared by adding pre-green dye The diode laser was irradiated immediately with 1 W, Exposure time of 10 s, 810 nm, continuous and non-contact mode.
  Other Names: Experimental: fluoride varinsh with laser application; Experimental: fluoride varnish without laser application
  Arms: fluoride varinsh with laser application; fluoride varnish without laser application

SUMMARY:
Dental caries is a very common condition, and although it has become less common, it still represents a serious public health risk. Caries symptoms range from the earliest molecular alterations in the tooth's apatite crystals to an apparent white spot lesion (WSL) or eventual cavitation. The white spot lesion looks chalky because minerals are being lost from both the surface and the underside of the enamel. A relatively simple and noninvasive caries preventive regimen in treating white spot lesions with low-level laser irradiation, either alone or with topical ﬂuoride treatment. This treatment results in reduced enamel solubility and dissolution.

DETAILED DESCRIPTION:
The study was reviewed and approved by the "Ethical research committee "of the Faculty of Dental Medicine for Girls; at Al-Azhar University, Cairo, Egypt. This study was conducted on 90 teeth with white spot lesions (WSLs) detected clinically on the buccal surface of teeth. The patients with WSLs were selected randomly from the operative dentistry clinic at the Faculty of Dentistry, Girl's Branch, Al-Azhar University

After examination, the teeth will be assigned into six groups of 15 teeth with white spot lesions each according to the remineralizing material used:

* The first group (A1B1): The teeth with WSL will be treated with nano-hydroxyapatite +fluoride with laser application.
* The second group (A1B2): The contralateral teeth will be treated with nano-hydroxyapatite +fluoride without laser application.
* The third group (A2B1): The teeth with WSL will be treated with nano-hydroxyapatite + xylitol with laser application.
* The fourth group (A2B2): The contralateral teeth will be treated with nano hydroxyapatite+ xylitol without laser application.
* The fifth group (A3B1): The teeth with WSL will be treated with 5% sodium fluoride varnish with laser application.
* The sixth group (A3B2): The contralateral teeth will be treated with 5% sodium fluoride without laser application.

ELIGIBILITY:
Inclusion Criteria:

* The patients should be 13-40 years old.
* Patients should have good oral hygiene.
* The patients with good general health and no systemic disease.

Exclusion Criteria:

* - Presence of enamel hypoplasia or dental fluorosis.
* Presence of carious cavity.
* Patients who have a significant medical history,
* Patients who have evidence of reduced salivary flow or significant tooth wear.

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — all selected patients were females for standardized in the study
Enrollment: 45 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Spectrophotometric color assessment: | from base line (application of materials) to one month
  The Vita Easy shade spectrophotometer (Vita Zahnfabrik, Bad Säckingen, Germany) was employed for the color assessment WSLs

SECONDARY OUTCOMES:
surface area measurement | from base line (application of materials) to one month
  after the finalization of the remineralization protocol, another radiographic examination was undertaken. Bitewing radiographs of the lesions were taken using the same X-ray unit, film holders for bite recording and vertical angulations for standardizing the geometric projection of the X-ray beam by digital subtraction radiograph.

CONTACTS AND LOCATIONS:
Overall Officials: Wael Essam, professor, Study Director — for Operative Dentistry Faculty of Dental Medicine for Girls Al-Azhar University
Locations (1):
- Al-Azhar University, Cairo, Egypt